CLINICAL TRIAL: NCT06622993
Title: Effectiveness of the SKILLS Program in the Management of Psychiatric Disorders: a Pilot Randomized Controlled Trial
Brief Title: Effectiveness of the SKILLS Program in the Management of Psychiatric Disorders
Acronym: P-SKILLS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DR240057
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Psychiatric Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Programm SKILLS (Experimental)
  Interventions: Other: Psychotherapy
- Waiting list (No Intervention)

INTERVENTIONS:
Other: Psychotherapy — The experimental group will receive the SKILLS program, i.e. 10 group psychotherapy sessions.
  Arms: Programm SKILLS

SUMMARY:
Epidemiological studies show that one person in eight suffers from at least one psychiatric disorder. Mental health is therefore a major public health issue, and care for these disorders must continue to be improved.

The management of mental disorders has long followed the traditional categorical approach of developing a treatment for a given disorder. However, researchers have recently pointed out the limits of this approach in the field of mental health. They highlight the large number of co-morbidities, the existence of aspecific disorders and the intra-diagnostic heterogeneity of patients. These factors have led them to develop a transdiagnostic approach, which focuses on the mechanisms common to the various disorders in order to treat them at the same time and thus reduce the cost of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Have at least one diagnosis of a psychiatric disorder
* Be able to carry out psychotherapy sessions
* Have been on stable psychiatric medication for 30 days
* Written informed consent obtained from the participant
* Be affiliated to a social security scheme or equivalent

Exclusion Criteria:

* Cognitive deficits marked by a score above the 10th percentile for one or more tests in the assessment history.
* Persons deprived of liberty by judicial or administrative decision; Persons under legal protection: guardianship or curatorship
* Presence of a severe depressive episode
* Be engaged in psychotherapeutic work elsewhere
* Presence of a state of excessive deficit, making psychotherapy impossible
* Presence of psychic decompensation (e.g. delusions) making psychotherapy impossible

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Evolution in Symptom Checklist Scale (SCL 90) scores between randomization and Month 3 | At the randomisation and Month 3

SECONDARY OUTCOMES:
Evolution of Transdiagnostic Skills Scale (T2S) score | At randomisation, Month 3 and Month 6
Evolution of Symptomatic Transdiagnostic Test (S2T) score | At randomisation, Month 3 and Month 6
Evolution of Hosptital Anxiety Depression Scalre (HADS) score | At randomisation, Month 3 and Month 6
Evolution of Satisfaction with Life Scale (SWLS) score | At randomisation, Month 3 and Month 6
Cumulative quantity of psychotropic treatment taken by patients (in mg) | At randomisation, Month 3 and Month 6